CLINICAL TRIAL: NCT01208298
Title: Study to Evaluate the Safety and Performance of Compeed® Cold Sore Patch Night in the Treatment of Herpes Labialis
Brief Title: Study to Evaluate Using a Cold Sore Patch to Treat Herpes Labialis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HCOWDH1001
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Herpes Labialis
Keywords: Cold Sore Patch
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- # 1727 (Experimental): Cold sore Patch
  Interventions: Device: Cold Sore Patch

INTERVENTIONS:
Device: Cold Sore Patch — All eligible subjects received CSP-Night at Screening Visit 1. Subjects were instructed to initiate therapy within approximately 1 hour of onset of their first sign or symptom. Treatment was continued until the lesion healed, or for a maximum of 10 days. All subjects were expected to return to the study center for clinical assessments within 24 hours and 48 hours after initiating treatment, and every other day thereafter, with a final visit at Day 10 or at the time of completion/ discontinuation if before Day 10.
  Other Names: Compeed® Cold Sore Patch Night

SUMMARY:
The primary objective of this study was to evaluate the safety and performance of a cold sore patch for the treatment of herpes labialis.

DETAILED DESCRIPTION:
This was an open, single-center multi-site, non-comparative study to evaluate the safety and performance of CSP-Night under actual-use conditions in subjects with herpes labialis of the lips and/or perioral skin. A sufficient number of subjects were screened to ensure that 45 subjects experienced and treated a cold sore outbreak in the course of 14 weeks. Subjects were instructed to initiate therapy within approximately 1 hour of onset of their first sign or symptom. Treatment was continued until the lesion healed, or for a maximum of 10 days. All subjects were expected to return to the study center for clinical assessments within 24 hours and 48 hours after initiating treatment, and every other day thereafter, with a final visit at Day 10 or at the time of completion/discontinuation if before Day 10. Diaries were completed each day, beginning upon initiation of therapy and continuing until study completion/ discontinuation, and included information on study product applications and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Females or males subjects, at least 18 to 70 years of age, in good general health
* History of recurrent herpes labialis (HSV-1) on the lips and/or perioral skin, with lesions typically manifesting as classical lesions (i.e., episodes progressing to vesicle, ulcer, and/or crust stages). Based on history, subject is considered likely to experience a cold sore outbreak within a time period of 2-3 months
* Individuals who were willing and able to provide informed consent
* Willing to stop all other treatment of this condition during the test period, including creams, tablets and other treatments
* Agrees not to use any topical product (e.g., cosmetics, lip balms, sunscreens) on the lesion area other than study medication
* Individuals who were willing to use the assigned test material for up to 10 consecutive days
* Individuals who were willing and able to follow the requirements for study participation
* Women of child bearing potential must agree to use an adequate method of birth control as defined by the protocol. Females who were post-menopausal (for at least 1 year), had a hysterectomy, bilateral ovariectomy or bilateral tubal ligation did not have to have additional birth control methods.

Exclusion Criteria:

* Individuals who were self reported to be pregnant, planning to become pregnant or nursing
* History of viral infection (e.g., hepatitis, HIV) or other condition likely to require treatment with systemic antiviral or steroid medications during the period of the study Note: Subjects suffering from chronic HSV and/ or have previously treated their herpes virus with systemic medication were permitted to be enrolled in this study.
* History of any malignant diseases
* Significant history of liver, kidney, heart, lung or digestive disease that required prolonged hospitalization or out-patient treatment
* Significant history of blood, nerve, brain or psychiatric disorders that required prolonged hospitalization or out-patient treatment
* Individuals with uncontrolled diabetes
* History of dermatologic or other condition(s) that in the judgment of the investigator may affect the course of the cold sore lesion or interfere with the actions of the study treatment or confound the interpretation of the study results
* Individuals using any analgesics or anti-inflammatory agents during the treatment period
* Individuals which were taking or had taken within the past 30 days of commencing treatment, systemic antiviral or steroid therapy
* Individuals which were taking or had taken within the past 7 days of commencing treatment, topical treatments for cold sore
* Individuals which were taking herbal supplements within 28 days of first dose of study product
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator
* Individuals with known sensitivity to any ingredients in the test product
* Individuals participating in another clinical research study, within 30 days of Visit 1 and at any time during the course of the treatment period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Clinician/Investigator's Global Assessment of Therapy | at discontinuation of therapy within 10 days
  Scores based on a on a scale from 0 = No response to therapy; 1 = Barely perceptible or minimal response to therapy; 2 = Very slight or low response to therapy; 3 = Slight or low response to therapy; 4 = Slight/low to moderate response to therapy; 5 = Moderate response to therapy; 6 = Moderate to substantial response to therapy; 7 = Substantial response to therapy; 8 = Substantial to significant response to therapy; 9 = Significant response to therapy; 10 = Excellent response to therapy
Subject's Global Assessment of Therapy | at discontinuation of therapy within 10 days
  Taking into account speed and quality of the response, subjects provided an overall assessment of the therapy with scores on a scale from 0= no response to 10= excellent response.

SECONDARY OUTCOMES:
Days to Heal | at day "healed" within 10 days
  Clinician/Investigator's assessed time to healing. The day the Clinician's assessment of lesion stage was "healed" was used as the time to heal score.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (2):
- United Kingdom (2):
  - 4 Front Research, Ellesmere Port, Cheshire
  - Intertek, Manchester, Manchester